CLINICAL TRIAL: NCT05595460
Title: Phase 1b Single Arm, Open-label Trial of RYZ101 in Combination With Carboplatin + Etoposide + Atezolizumab in Subjects With Somatostatin Receptor Expressing (SSTR+) Extensive Stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: Study of RYZ101 in Combination With SoC in Subjects With SSTR+ ES-SCLC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RayzeBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RYZ101-101
Record Dates: First submitted 2022-09-16; First posted 2022-10-27 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: SCLC,Extensive Stage
Keywords: actinium; alpha-emitter; SSTR+ ES-SCLC; SCLC; ES-SCLC; RYZ101; 225Ac; 225Ac-DOTATATE; targeted radiotherapy; atezolizumab; carboplatin; etoposide; radiopharmaceutical
MeSH Terms: interventions — atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RYZ101 + SoC (Experimental)
  Interventions: Drug: RYZ101 Dose Level 1; Drug: RYZ101 Dose Level 2; Drug: RYZ101 Dose Level 3; Drug: RYZ101 Dose Level -1; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: RYZ101 Dose Level 1 — Dose Level 1
Drug: RYZ101 Dose Level 2 — Dose Level 2
Drug: RYZ101 Dose Level 3 — Dose Level 3
Drug: RYZ101 Dose Level -1 — Dose Level -1
Drug: Atezolizumab — Atezolizumab
Drug: Carboplatin — Carboplatin
Drug: Etoposide — Etoposide

SUMMARY:
This study aims to determine the safety, preliminary antitumor activity, and pharmacokinetics (PK) of RYZ101 in combination with standard of care (SoC) therapy consisting of carboplatin + etoposide + atezolizumab in untreated subjects with somatostatin receptor expressing (SSTR+) ES-SCLC.

ELIGIBILITY:
INCLUSION CRITERIA

* Age of at least 18 years at the time of signing the informed consent.
* Cytologically or histologically confirmed ES-SCLC (American Joint Committee on Cancer [AJCC] 8th edition) and is untreated or received ≤1 cycle of platinum-etoposide and PD-L1 inhibitor therapy. It is acceptable to omit the first dose of PD-L1 inhibitor therapy due to logistical reasons if receiving SoC during or prior to the start of the screening period.
* Subject is a candidate for therapy with SoC which includes:

  * Carboplatin for a maximum of 4 cycles
  * Etoposide for a maximum of 4 cycles
  * Atezolizumab
* At least 1SSTR-PET imaging-positive measurable site of disease (according to RECIST v1.1) and ≥50% of RECIST v1.1 measurable metastatic lesions must be SSTR-imaging positive.
* Adequate hematologic, renal and hepatic function

EXCLUSION CRITERIA

* Prior exposure to immune-mediated therapy,
* Known active or suspected autoimmune disease or any condition requiring systemic treatment with immunosuppressive medications within 14 days prior to first dose of study drug
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis. Note: History of radiation pneumonitis is permitted.
* Severe infection within 4 weeks and/or treatment with therapeutic oral or i.v. antibiotics within 2 weeks prior to initiation of study treatment.
* Prior allogeneic stem cell or solid organ transplantation.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab.
* Radiotherapy to the chest prior to systemic therapy or planned consolidation chest radiation therapy. Radiation therapy outside of the chest for palliative care is allowed but must be completed >2 weeks prior to first dose of study drug.
* Significant cardiovascular disease and/or resistant hypertension
* Subjects with previously treated central nervous system (CNS) metastases who have not recovered from acute side effects of radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
RP2D | 42 days of study treatment
  RP2D as determined by incidence rate of DLTs
Safety and tolerability of RYZ101 in combination with SoC | Up to 50 months
  Safety and tolerability of RYZ101 in combination with SoC as measured by incidence and severity of AEs including SAEs, laboratory changes and other safety findings

CONTACTS AND LOCATIONS:
Overall Officials: Petrus De Jong, MD, Study Director — RayzeBio, Inc.
Locations (15):
- United States (14):
  - Research Facility, Los Angeles, California
  - Research Facility, San Francisco, California
  - Research Facility, Jacksonville, Florida
  - Research Facility, Miami, Florida
  - Research Facility, Orlando, Florida
  - Research Facility, Iowa City, Iowa
  - Reserach Facility, Lexington, Kentucky
  - Research Facility, Grand Rapids, Michigan
  - Research Facility, Troy, Michigan
  - Research Facility, Rochester, Minnesota
  - Research Facility, St Louis, Missouri
  - Research Facility, Omaha, Nebraska
  - Research Facility, Houston, Texas
  - Research Facility, Salt Lake City, Utah
- Research Facility, San Juan, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: No